CLINICAL TRIAL: NCT05465577
Title: Coverage and Cost-of-Care Links Financial Navigation Program in Hematology and Blood and Bone Marrow Transplantation (BMT)
Brief Title: Coverage and Cost-of-Care (CC) Links- Financial Navigation Program
Acronym: CC Links
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jean Edward (Other)
Responsible Party: Sponsor-Investigator, Jean Edward, Associate Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MCC-20-61653
Record Dates: First submitted 2022-07-15; First posted 2022-07-20 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Financial Stress; Hematologic Cancer; Survivorship
Keywords: financial navigation; quality of life; hardship; caregivers; financial toxicity
MeSH Terms: conditions — Financial Stress; Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Financial Navigation- Patients Only (Experimental): Patients only participated in financial navigation program.
  Interventions: Other: CC Links
- Financial Navigation- Patient and Caregiver (Experimental): Patients and their caregivers participated as a dyad in financial navigation program.
  Interventions: Other: CC Links

INTERVENTIONS:
Other: CC Links — The CC Links intervention is built on a platform of interdisciplinary team-based science, which ensured that the financial navigator worked closely with other members of the healthcare team including oncologists, nurses, transplant coordinators, social workers, and case managers, to help enhance financial hardship screening and connect survivors and caregivers with financial assistance services.

SUMMARY:
This trial is a mixed-methods, non-randomized design guided by the Consolidated Framework for Implementation Research (CFIR) to develop, implement, and evaluate Coverage and Cost-of-Care Links (CC Links) -a novel financial navigation intervention for hematologic cancer survivors and their caregivers.

DETAILED DESCRIPTION:
The CC Links intervention included an oncology financial navigator who worked in the Hematology-Oncology Clinic. The navigator's functions included: screening for financial hardship to identify unmet financial needs (using the Comprehensive Score for Financial Toxicity (COST) and National Comprehensive Cancer Network's Distress Thermometer; initiating cost of care conversations; providing cost of care estimates; ensuring adequate health insurance coverage and assisting with applying for additional coverage; assisting with internal financial assistance program applications; connecting survivors/caregivers with disease specific resources and other external assistance programs; coordinating discharge planning; referring survivors to social workers and other staff/resources as needed; and, coordinating financial assistance services as survivors/caregivers transition between outpatient and inpatient settings.

ELIGIBILITY:
Inclusion Criteria:

* hematological cancer patients from the Division of Hematology and Bone Marrow Transplantation at the University of Kentucky
* caregivers of cancer patients
* positive screening for financial hardship

Exclusion Criteria:

- unable to provide consent

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Change in coping behaviors | Approximately 8 months (baseline and following resolution of financial needs)
  "Coping behaviors" was measured using a series of 9 yes/no items that first assess whether any recommended cancer care was skipped for any reason (yes/no), and then whether the reason for not receiving the care that they or their doctor believed necessary was due to any of 8 listed reasons (yes/no for each). Typical reasons included 'Couldn't afford care,' 'Insurance company wouldn't approve or pay for care,' and 'Had problems getting to the doctor's office.' The sum of the number of yes responses is the total score, with higher scores indicating greater coping behaviors in response to financial hardship. The items in this scale are from the Medical Expenditure Panel Survey - Experiences with Cancer Survivorship Survey (MEPS-ECSS).
Change in material conditions | Approximately 8 months (baseline and following resolution of financial needs)
  "Material conditions" was measured using 8 items (6 from the Medical Expenditure Panel Survey: Experiences with Cancer Survivorship Supplement (MEPS-ECSS) and 2 from demographic survey) that measure the financial condition of the participant with cancer and their family. Six of the items are yes/no and these include questions on borrowing money or go into debt, filing for bankruptcy, and concerns about having to pay large medical bills because of the cost of cancer treatment. The remaining two items are ordinal and measure the amount of debt related to cancer costs (options range from $0 to $100,00+), and the how they perceive their household's income currently (choices range from 'living comfortably on present income' to 'finding it very difficult on present income'). The latter two items are rescaled to 0-1 variables, so they have the same ranges as the yes/no items and are summed to create the total score. Higher scores indicate greater financial hardship.
Change in psychological response (financial toxicity) | Approximately 8 months (baseline and following resolution of financial needs)
  Psychological response (i.e. financial toxicity) was measured using the 11-item Comprehensive Score for Financial Toxicity (COST) that measures emotional aspects of financial hardship (financial toxicity) among cancer patients. Each item is scored on a 5-point ordinal scale ranging from 0='Not at all' to 4='Very much.' Sample items include 'My out-of-pocket expense are more than I thought they would be' and 'I am frustrated that I cannot work or contribute as much as I usually do.' Lower values indicate greater financial toxicity.
Change in health-related quality of life | Approximately 8 months (baseline and following resolution of financial needs)
  Health-related QOL was measured using four Patient-Reported Outcomes Measurement Information System (PROMIS) scales.xx Each of these were scored and standardized by submitting the raw values to the HealthMeasures scoring service. standardized values of the total scores were used throughout the analysis for this study. The four scales include the PROMIS physical health and emotional health subscales (from the 10-item PROMIS Scale v1.2 - Global Health),xx the 4-item PROMIS- Anxiety Short Form, and the 6-item PROMIS-Depression Short Form. The physical (physical health, function, pain, and fatigue items) and emotional health (QOL, mental health, social activities, and emotional problem items) subscales are each based on 4 items, with higher scores indicating a more positive health self-assessment. For the anxiety and depression scales, higher scores indicate a greater manifestation of symptoms.
Change in distress. | Approximately 8 months (baseline and following resolution of financial needs)
  Distress was measured using the National Comprehensive Cancer Network's (NCCN) Distress Thermometer and its accompanying 40-item problem list. A cutoff score of 4 indicated clinically elevated distress levels

SECONDARY OUTCOMES:
Financial Savings | Approximately at 8 months (following resolution of financial needs)
  Amount of money saved per patient including grants and financial assistance received, total charges, financial assistance adjustments, insurance payments, and insurance charges.

CONTACTS AND LOCATIONS:
Overall Officials: Jean S Edward, PhD, RN, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No